CLINICAL TRIAL: NCT03454594
Title: Laser Hemotherapy Trial for Coronary Artery Disease Prevention in High Risk Patients
Brief Title: Watch Laser Acupuncture With Nasal Radiation for Prevention of Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ebtesam Nabil, lecturer assistance at Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/001561
Record Dates: First submitted 2018-02-25; First posted 2018-03-06 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Cardiovascular Risk Factor; Coronary Artery Disease
Keywords: hypertension; high blood viscosity; hypercholesterolemia
MeSH Terms: conditions — Coronary Artery Disease; Hypertension; Hypercholesterolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low level laser hemotherapy (Experimental): Watch laser acupuncture and nasal irradiation
  Interventions: Device: low level laser hemotherapy
- control (No Intervention): all the participants in this group did not receive low level laser irradiation during the study period

INTERVENTIONS:
Device: low level laser hemotherapy — semiconductor laser therapeutic instrument irradiate the circulating blood in the vessels of left hand acupoint and the mucosal tissue in the nasal cavity
  Other Names: Watch laser
  Arms: low level laser hemotherapy

SUMMARY:
This study will evaluate the effect of low level laser blood radiation applied to all participants for prevention of coronary artery disease in patients with high risk (hypertension,high blood viscosity, hypercholesterolemia as well as related immune issues)

DETAILED DESCRIPTION:
The areas of low - intensity laser use have expanded in several conditions by different mechanisms and ways. Hypertension as one of coronary artery disease risk factors and early indicator of future cardiovascular events with high blood viscosity and elevated blood cholesterol levels with immune-pathological basis became necessary issue to be handled. Low Level Laser irradiation effects on blood is very essential way in revealing the mechanisms of the action of laser radiation on biological tissues by means of changes in metabolism, leading to molecular, cellular and systemic changes.

ELIGIBILITY:
Inclusion Criteria:

* stage I hypertensive patients
* patients from 30 to 34.9 kg/m2 body mass index
* medically stable patients
* all participants have sufficient cognition enough to understand the requirements of the study

Exclusion Criteria:

* history of malignant disease
* smoking
* history of progressive fatal disease
* history of drug or alcohol abuse
* blood donation within at least 30 days
* pregnant, trying to be pregnant or breast feeding
* cognitive impairment that will make it difficult to partake in the study

Ages: 55 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-08-05 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
changes of blood pressure | 8 weeks
  measuring blood pressure before and after each low level laser radiation

SECONDARY OUTCOMES:
changes in blood viscosity | 8 weeks
  measuring changes in blood viscosity before and after low level laser radiation session
change in IL-17 level | 45 days
  measuring changes in IL-17 level before and after low level laser radiation session
change in functional capacity | 70 days
  measuring of 6 minute walking test before and after low level laser irradiation as an indicator of functional capacity improving
change in CD 8 (cluster of differentiation 8) level | 45 days
  measuring changes in CD 8 (cluster of differentiation 8) level before and after low level laser radiation session
change in TC (total cholesterol) level | 60 days
  measuring changes in TC (total cholesterol) level before and after low level laser radiation session
change in LDL (low density lipoprotien) level | 60 days
  measuring changes in LDL (low density lipoprotien) level before and after low level laser radiation session
change in TG (triglyceride) level | 60 days
  measuring changes in TG (triglyceride) level before and after low level laser radiation session
change in HDL (high density lipoprotien) level | 60 days
  measuring changes in HDL (high density lipoprotien) level before and after low level laser radiation session

CONTACTS AND LOCATIONS:
Overall Officials: Cairo Giza, MD, Principal Investigator — Cairo University
Locations (1):
- Cairo, Giza, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: Yes
De-identified participated data for underlie results reported in this trial
Supporting Information: Study Protocol
Time Frame: data will be available after 6 months of study completion and ending 36 months
Access Criteria: proposals should directed to Dr.EbtesamNagy@cu.edu.eg. To gain access, data requestors will need to sign a data access agreement